CLINICAL TRIAL: NCT04878900
Title: EVALUATION OF THE EFFECTS OF THE COVID-19 PANDEMIC ON PAIN, STRESS, SLEEP AND QUALITY OF LIFE IN PATIENTS WITH CHRONIC MUSCULOSKELETAL PAIN
Brief Title: Effects of COVID-19 in Chronic Pain
Status: Completed | Type: Observational
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Elzem Bolkan Günaydın, Principal investigator, Ufuk University
Other Study IDs: 2020-3-16
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Chronic Pain; Covid19
MeSH Terms: conditions — Chronic Pain; COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Survey

SUMMARY:
The aim of this study is to evaluate the effects of the COVID-19 pandemic on pain, stress, sleep and quality of life in patients with chronic musculoskeletal pain and the relationships between them. In this cross-sectional study, 100 volunteer patients aged 18-65 years with chronic (longer than 3 months) musculoskeletal pain were included. Age, gender, body-mass index (BMI) and systemic diseases of the participants were recorded as demographic data. Data were collected regarding the area of the body where pain is most dominant in the musculoskeletal system and how long the pain has been in these area, whether there is routine use of analgesics before and after the pandemic and the amount if any, whether the person or the person's relatives have a history of COVID-19, whether exercising regularly before and after the pandemic. Afterwards, the participants were asked to evaluate their general pain severity and global well-being assesment with the visual analog scale (VAS) in the pre-pandemic period and in the last month. For pain severity, the patients marked their pain severity on a line of 10 centimeters (cm) with the starting point (0) expressing no pain, and the end point (10) expressing the most severe pain experienced in life; for patient's global assesment the patients marked their global assesment on a line of 10 centimeters (cm) with the starting point (0) expressing very good, and the end point (10) expressing very bad. The distance between the point marked by the patient and the starting point was measured. The higher the measured value meant the greater the severity of the patient's pain and the worse the patient's global assessment [11]. Subsequently, the patients were asked to answer questions on the Perceived Stress Scale (PSS), Pittsburgh Sleep Quality Index (PSQI) and Nottingham Health Profile (NHP) scales.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years with chronic (longer than 3 months) musculoskeletal pain

Exclusion Criteria:

* Having a history of trauma and surgical intervention in the last 3 months,
* Having a history of known inflammatory rheumatic disease,
* Having a history of chronic severe systemic or neurological disease,
* Having a moderate or severe impairment of cognitive status determined by the minimental test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 years with chronic (longer than 3 months) musculoskeletal pain
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
General pain severity and global well-being assesment with the visual analog scale (VAS). | 2 months
  For pain severity, the patients marked their pain severity on a line of 10 centimeters (cm) with the starting point (0) expressing no pain, and the end point (10) expressing the most severe pain experienced in life; for patient's global assesment the patients marked their global assesment on a line of 10 centimeters (cm) with the starting point (0) expressing very good, and the end point (10) expressing very bad.
Perceived Stress Scale (PSS) | 2 months
  It is a scale to evaluate how stressful some situations in life are perceived by the individual. The long form of the scale consists of 14 items in total. The situations given in each item are evaluated with a 5-point Likert-type scale (0=never, 1=almost never, 2=sometimes, 3=fairly often, 4=very often). The scale has two short forms consisting of 10 and 4 items. The total score ranges from 0-56 for PSS-14, 0-40 for PSS-10, and 0-16 for PSS-4. The higher the scores, the greater the person's perception of stress.
Pittsburgh Sleep Quality Index (PSQI) | 2 months
  It is a scale to evaluate sleep quality and disorders. It consists of 24 questions in total. 19 questions are self-assessment questions, 5 questions are assessment questions made by their spouse or roommate. 18 question items are used in scoring. The scale consists of 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medication, and daytime dysfunction. While some of the components consist of a single question item, some are formed by grouping several items. Each component is scored between 0 and 3 points, and the total score of the components gives the total score of the scale. The higher the total score the worse the sleep quality.
Nottingham Health Profile (NHP) | 2 months
  It is a general health status scale that evaluates perceived problems in physical, emotional and social areas and how these problems affect daily activities. The questions in the first part of the scale are about the health status of the people, and the questions in the second part are about the effects of their health status on daily life. The first part consists of 38 items in which each item is answered as yes or no. This section has a total of 6 sub-dimensions: pain, emotional reactions, sleep, social isolation and physical mobility and energy. The higher the score, the worse the perception of quality of life regarding health status. The second part consists of 7 items that question whether there are problems in the daily life areas that are most likely to be affected by the health condition of the person, such as work life, housework, social life, interpersonal relationships, sexual life, hobbies and holidays, each item being answered as yes or no.

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No